CLINICAL TRIAL: NCT04164251
Title: Inpatient Screening Mammography for Non-adherent and High Risk Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Maryland Cigarette Restitution Fund (Other Government); EQUIP (Excellence in Quality, Utilization of resources, Integration and Patient- centered Care) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: NA_00079826
Record Dates: First submitted 2019-11-12; First posted 2019-11-15 (Actual); Last update posted 2019-12-03 (Actual); Status verified 2019-11

CONDITIONS: Breast Cancer
Keywords: Breast Cancer Screening; Mammography
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Inpatient screening mammography for non-adherent and high risk (Experimental): All non-adherent women were offered inpatient screening mammography during hospitalization
  Interventions: Other: Screening mammography

INTERVENTIONS:
Other: Screening mammography — The purpose of the study was to evaluate the feasibility of securing inpatient breast cancer screening mammograms for non-adherent hospitalized women prior to hospital discharge.

SUMMARY:
The investigators propose to pilot a program that will evaluate the feasibility of an inpatient screening mammography for non-adherent and high risk hospitalized women age 52-74 admitted to the medicine services at Johns Hopkins Bayview Medical Center and Howard County General Hospital. The two key activities include: inpatient breast care education with educational handouts and offering inpatient screening mammography. Inpatient screening mammography will be offered to non-adherent (last screening mammogram more than 24 months ago) and high risk (Gail 5-year risk of breast cancer 1.6 or greater) women. This pilot program will thus evaluate the feasibility of an inpatient screening mammography as an innovative approach to increase breast cancer screening among non-adherent and high risk women.

ELIGIBILITY:
Inclusion Criteria:

* women between 50 and 74 years of age who were non-adherent to breast screening guidelines

Exclusion Criteria:

* Patients with a history of breast cancer or mastectomy
* history of other cancers (except skin)
* serious comorbidities making patient's life expectancy <10 years

Ages: 50 Years to 74 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — women between 50 and 74 years of age who were non-adherent to breast screening guidelines (USPSTF recommendations)
Enrollment: 101 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Proportion of women who underwent a screening mammography during hospitalization | Prior to hospital discharge, up to 1 year
  Screening mammography is done during hospitalization. Proportion of women that get the screening will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Waseem Khaliq, MD, Principal Investigator — Johns Hopkins University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Khaliq W, Siferd C, Kantsiper ME, Jacobs L, Howell EE, Wright SM. Capturing the Rest: Inpatient Mammography for Nonadherent Hospitalized Women. Am J Prev Med. 2021 Nov;61(5):709-715. doi: 10.1016/j.amepre.2021.04.026. Epub 2021 Jul 4. PMID 34229929